CLINICAL TRIAL: NCT01700140
Title: Phase II Clinical Study of SyB D-0701 for Radiotherapy Induced Nausea and Vomiting
Brief Title: Phase II Study of SyB D-0701 for Radiotherapy-Induced Nausea and Vomiting (RINV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: Double
Other Study IDs: 2010003
Record Dates: First submitted 2012-09-11; First posted 2012-10-04 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Radiotherapy-induced Nausea and Vomiting (RINV)
MeSH Terms: conditions — Vomiting

ARMS (3):
- SyB D-0701: high dose group (Experimental)
  Interventions: Drug: SyB D-0701
- SyB D-0701: low dose group (Experimental)
  Interventions: Drug: SyB D-0701; Drug: Placebo
- placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SyB D-0701 — Study drug patches [Low dose group (18.75 mg): SyB D-0701 15 cm2 placebo patch + SyB D-0701 25 cm2 patch, High dose group (30.00 mg): SyB D-0701 15 cm2 patch + SyB D-0701 25 cm2 patch] assigned at the Case Registration Center are applied to either the right or left upper arm at 12 to 24 hours prior to the start of radiotherapy and left as is until 24 hours after completion of the third irradiation.
  Arms: SyB D-0701: high dose group; SyB D-0701: low dose group
Drug: Placebo — Study drug patches (Placebo group: SyB D-0701 15 cm2 placebo patch + SyB D-0701 25 cm2 placebo patch) assigned at the Case Registration Center are applied to either the right or left upper arm at 12 to 24 hours prior to the start of radiotherapy and left as is until 24 hours after completion of the third irradiation.
  Arms: SyB D-0701: low dose group; placebo group

SUMMARY:
The purpose of this study is to explore the dose response of SyB D-0701 for preventing nausea and emesis associated with radiotherapy (fractionated/localized irradiation) in cancer patients scheduled to receive radiotherapy (fractionated/localized irradiation) alone.

DETAILED DESCRIPTION:
Exploratory study of dose response of SyB D-0701 to preventing effects for nausea and emesis associated with radiotherapy (fractionated/localized irradiation)

ELIGIBILITY:
Inclusion Criteria Patients must satisfy the following conditions listed below.

1. Patients with histologically verified malignant tumors
2. Patients receiving radiotherapy alone who are scheduled for at least 3 fractions, each at a radiation dose of 1.5 to 3.0 Gy
3. Cancer patients scheduled for radiotherapy over a field of at least 100 cm2 (50 cm2 or more in cases of irradiation of the vertebrae only) that includes the abdomen and pelvis (region with upper edge at the 11th thoracic vertebrae and lower edge at pelvic cavity)
4. Patients not scheduled to receive anti-tumor agents between the first and the fifth day of radiotherapy. If the patient has a history of anti-tumor agent therapy, however, at the time of the patient's registration, at least 5 days must have elapsed since drug administration was terminated, and the patient must not be scheduled to receive any anti-tumor agent from the first to the fifth day of radiotherapy
5. Male patients who are surgically sterilized, or who agree to practice adequate contraception during the study
6. Female patients of child-bearing potential who agree to practice adequate contraception during the study
7. Patients whose performance status (PS) of Eastern Cooperative Oncology Group (ECOG) is 0 to 2
8. Patients who were at least 20 years of age when their consent was obtained
9. Patients who have given consent in writing to participate in the study with full understanding of the explanatory documents

Exclusion Criteria Patients who satisfy any of the following conditions will not be enrolled in the study.

1. Patients with nausea and/or emesis; patients who also have intestinal obstruction, vestibular dysfunction (e.g., epilepsy), Meniere's syndrome, cerebral metastasis, electrolyte imbalance (hypercalcemia, hyperglycemia, hyponatremia), uremia, etc., and patients for whom it is judged that there is a high probability that their nausea or emesis arises from the aforementioned causes. Registration is possible, however, for patients with motion sickness (vehicle sickness) or patients with temporary nausea/emesis arising from routine activities.
2. Patients with primary or metastasized brain tumors who show signs of elevated intracranial pressure
3. Patients who previously received radiotherapy to the brain or to the region that includes the abdomen and pelvis (region with upper edge at the 11th thoracic vertebrae and lower edge at pelvic cavity)
4. Patients who take drugs that affect the evaluation of nausea or emesis (rescue medication and 5-hydroxytryptamine 3 (5-HT3) receptor antagonists, neurokinin 1 (NK1) receptor antagonists, anxiolytics, psychotropic drug, opioid analgesics and corticosteroid [systemic administration] except for rescue medication)
5. Patients with abnormal findings (e.g., erythema, rash, wounds) at sites where the study drug has been applied
6. Patients with a history of hypersensitivity to study drug ingredients or to other 5-HT3 receptor antagonists
7. Patients with a history of allergy involving dermal symptoms
8. Patients with clear signs of infection (including viral infection)
9. Patients with complications from drug or alcohol dependence, or with a history of the same
10. Patients who have participated in some type of clinical study (including physician-initiated clinical studies or clinical research) within 3 months prior to their registration for the present study and who have been given a study drug (including drugs not yet approved). Patients can be registered for this study, however, if they have participated in a clinical study, etc., in which only drugs already approved have been used.
11. Patients with serious hepatic or renal damage [Grade 3 or above in the Common Terminology Criteria for Adverse Events (CTCAE) (ver. 4.0-JCOG)]
12. Patients with cardiac dysfunction
13. Patients who are pregnant, who might be pregnant or who are currently lactating
14. Other patients judged as unsuitable by the investigator or sub-investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- Japan (21):
  - Research site, Nagoya, Aichi-ken
  - Research site, Kashiwa, Chiba
  - Research site, Matsuyama, Ehime
  - Research site, Kurume, Fukuoka
  - Research site, Maebashi, Gunma
  - Research site, Ōta, Gunma
  - Research site, Hiroshima, Hiroshima
  - Research site, Sapporo, Hokkaido
  - Research site, Sagamihara, Kanagawa
  - Research site, Yokohama, Kanagawa
  - Research, Kyoto, Kyoto
  - Research site, Kashihara, Nara
  - Research site, Niigata, Niigata
  - Research site, Nakagami, Okinawa
  - Research site, Sayama, Osaka
  - Research site, Hidaka, Saitama
  - Research site, Kitaadachi, Saitama
  - Research Site, Koshigaya, Saitama
  - Reseach site, Tokyo, Tokyo
  - Research site, Tokyo, Tokyo
  - Research site, Yamagata, Yamagata

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group: Study drug patches (Placebo group: SyB D-0701 15 cm2 placebo patch + SyB D-0701 25 cm2 placebo patch) assigned at the Case Registration Center are applied to either the right or left upper arm at 12 to 24 hours prior to the start of radiotherapy and left as is until 24 hours after completion of the third irradiation.
- SyB D-0701: Low Dose Group: Study drug patches [Low dose group (18.75 mg): SyB D-0701 15 cm2 placebo patch + SyB D-0701 25 cm2 patch (18.75 mg)] assigned at the Case Registration Center are applied to either the right or left upper arm at 12 to 24 hours prior to the start of radiotherapy and left as is until 24 hours after completion of the third irradiation.
- SyB D-0701: High Dose Group: Study drug patches [High dose group (30.00 mg): SyB D-0701 15 cm2 patch (11.25 mg) + SyB D-0701 25 cm2 patch (18.75 mg)] assigned at the Case Registration Center are applied to either the right or left upper arm at 12 to 24 hours prior to the start of radiotherapy and left as is until 24 hours after completion of the third irradiation.
Period: Overall Study
Arm/Group | Placebo Group | SyB D-0701: Low Dose Group | SyB D-0701: High Dose Group
Started | 61 | 66 | 62
Completed | 55 | 57 | 61
Not Completed | 6 | 9 | 1
Not completed — Use of rescue drugs | 3 | 3 | 1
Not completed — Discontinuation of radiotherapy | 1 | 0 | 0
Not completed — Use of chemotherapy or surgical therapy | 0 | 1 | 0
Not completed — Aggravation of symptoms | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Inclusion/exclusion criteria deviation | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Per protocol set:
  Of all the randomized subjects, those who were compliant with the protocol were included in the per protocol set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | SyB D-0701: Low Dose Group | SyB D-0701: High Dose Group | Total
Number analyzed (Participants) | 56 | 59 | 60 | 175
Age, Customized [Number; unit: Participants]
  20-40 years | 3 | 7 | 3 | 13
  40-50 years | 11 | 8 | 7 | 26
  50-60 years | 11 | 13 | 17 | 41
  60-70 years | 14 | 14 | 12 | 40
  70≤ years | 17 | 17 | 21 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 35 | 35 | 108
  Male | 18 | 24 | 25 | 67
Metastasis [Number; unit: Participants]
  Absent | 32 | 24 | 36 | 92
  Present | 24 | 35 | 24 | 83
History of radiotherapy [Number; unit: Participants]
  Absent | 53 | 54 | 60 | 167
  Present | 3 | 5 | 0 | 8
History of recent chemotherapy [Number; unit: Participants]
  Absent | 37 | 36 | 38 | 111
  Present | 19 | 23 | 22 | 64
Complication [Number; unit: Participants]
  Absent | 2 | 11 | 10 | 23
  Present | 54 | 48 | 50 | 152
Diseases in the past 5 years [Number; unit: Participants]
  Absent | 23 | 29 | 22 | 74
  Present | 33 | 30 | 38 | 101
History of smoking habit [Number; unit: Participants]
  Absent | 29 | 31 | 39 | 99
  Present | 27 | 28 | 21 | 76
Alcohol consumption history [Number; unit: Participants]
  Absent | 36 | 32 | 40 | 108
  Present | 20 | 27 | 20 | 67
Motion sickness (vehicle sickness) [Number; unit: Participants]
  Absent | 54 | 57 | 55 | 166
  Present | 2 | 2 | 5 | 9
Performance status [Number; unit: Participants] — The criteria of Eastern Cooperative Oncology Group (ECOG) performance status are shown below.
  0: Fully active, able to carry on all pre-disease performance without restriction, 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2: Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  Participants
    0 | 39 | 41 | 50 | 130
    1 | 14 | 16 | 8 | 38
    2 | 3 | 2 | 2 | 7
Nausea/emesis [Number; unit: Participants]
  Absent | 56 | 59 | 60 | 175
  Present | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Complete Control (no Signs of Emesis or Moderate to Severe Nausea and no Use of Rescue Medication) Rate From the Start of Radiotherapy Until 24 Hours After the Third Irradiation
Description: The complete control rate was defined as the percentage of subjects who had no emesis and no moderate or more severe nausea and who used no rescue drugs during the period from the time of the first irradiation to 24 hours after the third irradiation.
Time Frame: 72 hours
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Group | SyB D-0701: Low Dose Group | SyB D-0701: High Dose Group
Number analyzed (Participants) | 56 | 59 | 60
Percentage of participants | 85.7 | 84.7 | 93.3
Statistical Analysis 1: Comparison: Placebo Group vs SyB D-0701: Low Dose Group; Test type: Superiority or Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Placebo Group vs SyB D-0701: High Dose Group; Test type: Superiority or Other; p = 0.2284, Fisher Exact
Statistical Analysis 3: Comparison: Placebo Group vs SyB D-0701: Low Dose Group vs SyB D-0701: High Dose Group; Test type: Superiority or Other; p = 0.2549, Cochran-Armitage test

2. Secondary Outcome: Complete Response (no Signs of Emesis and no Use of Rescue Medication) Rate From the Start of Radiotherapy Until 24 Hours After the Third Irradiation
Description: The complete response rate was defined as the percentage of subjects who had no emesis and who used no rescue drugs during the period from the time of the first irradiation to 24 hours after the third irradiation.
Time Frame: 72 hours
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Group | SyB D-0701: Low Dose Group | SyB D-0701: High Dose Group
Number analyzed (Participants) | 56 | 59 | 60
Percentage of participants | 89.3 | 88.1 | 96.7
Statistical Analysis 1: Comparison: Placebo Group vs SyB D-0701: Low Dose Group; Test type: Superiority or Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Placebo Group vs SyB D-0701: High Dose Group; Test type: Superiority or Other; p = 0.1527, Fisher Exact
Statistical Analysis 3: Comparison: Placebo Group vs SyB D-0701: Low Dose Group vs SyB D-0701: High Dose Group; Test type: Superiority or Other; p = 0.1864, Cochran-Armitage test

3. Secondary Outcome: Time to First Emesis
Description: Time from the start of radiotherapy to the onset of first emesis. The median (50% point) of time to first emesis was estimated.
Time Frame: 24-72 hours
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Placebo Group | SyB D-0701: Low Dose Group | SyB D-0701: High Dose Group
Number analyzed (Participants) | 56 | 59 | 60
Hours | NA [NA to NA] — The estimated non-incidence of emesis by the Kaplan-Meier method exceeded 50%. | NA [NA to NA] — The estimated non-incidence of emesis by the Kaplan-Meier method exceeded 50%. | NA [NA to NA] — The estimated non-incidence of emesis by the Kaplan-Meier method exceeded 50%.
Statistical Analysis 1: Comparison: Placebo Group vs SyB D-0701: Low Dose Group; Test type: Superiority or Other; p = 0.8361, Generalized Wilcoxon test; Hazard Ratio (HR) = 0.918, 95% CI 2-sided [0.266 to 3.172]
Statistical Analysis 2: Comparison: Placebo Group vs SyB D-0701: High Dose Group; Test type: Superiority or Other; p = 0.0724, Generalized Wilcoxon test; Hazard Ratio (HR) = 0.423, 95% CI 2-sided [0.144 to 1.237]

4. Secondary Outcome: Time to First Nausea
Description: Time from the start of radiotherapy to the onset of first nausea. The median (50% point) of time to first nausea was estimated.
Time Frame: 24-72 hours
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Placebo Group | SyB D-0701: Low Dose Group | SyB D-0701: High Dose Group
Number analyzed (Participants) | 56 | 59 | 60
Hours | NA [NA to NA] — The estimated non-incidence of nausea by the Kaplan-Meier method exceeded 50%. | NA [NA to NA] — The estimated non-incidence of nausea by the Kaplan-Meier method exceeded 50%. | NA [NA to NA] — The estimated non-incidence of nausea by the Kaplan-Meier method exceeded 50%.
Statistical Analysis 1: Comparison: Placebo Group vs SyB D-0701: Low Dose Group; Test type: Superiority or Other; p = 0.6466, Generalized Wilcoxon test; Hazard Ratio (HR) = 1.213, 95% CI 2-sided [0.616 to 2.388]
Statistical Analysis 2: Comparison: Placebo Group vs SyB D-0701: High Dose Group; Test type: Superiority or Other; p = 0.2701, Generalized Wilcoxon test; Hazard Ratio (HR) = 0.828, 95% CI 2-sided [0.566 to 1.210]

5. Secondary Outcome: Complete Control Rate Within 24 Hours After Each Irradiation From Sessions 1 to 3
Description: Complete control rate within 24 hours after each irradiation, from the first to the third fraction of radiotherapy.
  The complete control rate was defined as the percentage of subjects who had no emesis and no moderate or more severe nausea and who used no rescue drugs.
Time Frame: 24-72 hours
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Group | SyB D-0701: Low Dose Group | SyB D-0701: High Dose Group
Number analyzed (Participants) | 56 | 59 | 60
Percentage of participants
  First irradiation | 91.1 | 89.8 | 98.3
  Second irradiation | 90.9 | 94.7 | 98.3
  Third irradiation | 89.1 | 96.4 | 94.9
Statistical Analysis 1: Comparison: Placebo Group vs SyB D-0701: Low Dose Group; Statistical analysis for complete control rate after the first irradiation; Test type: Superiority or Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Placebo Group vs SyB D-0701: High Dose Group; Statistical analysis for complete control rate after the first irradiation; Test type: Superiority or Other; p = 0.1051, Fisher Exact
Statistical Analysis 3: Comparison: Placebo Group vs SyB D-0701: Low Dose Group; Statistical analysis for complete control rate after the second irradiation; Test type: Superiority or Other; p = 0.4856, Fisher Exact
Statistical Analysis 4: Comparison: Placebo Group vs SyB D-0701: High Dose Group; Statistical analysis for complete control rate after the second irradiation; Test type: Superiority or Other; p = 0.1047, Fisher Exact
Statistical Analysis 5: Comparison: Placebo Group vs SyB D-0701: Low Dose Group; Statistical analysis for complete control rate after the third irradiation; Test type: Superiority or Other; p = 0.1617, Fisher Exact
Statistical Analysis 6: Comparison: Placebo Group vs SyB D-0701: High Dose Group; Statistical analysis for complete control rate after the third irradiation; Test type: Superiority or Other; p = 0.3099, Fisher Exact

6. Secondary Outcome: Complete Response Rate Within 24 Hours After Each Irradiation From Sessions 1 to 3
Description: Complete response rate within 24 hours after each irradiation, from the first to the third fraction of radiotherapy.
  The complete response rate was defined as the percentage of subjects who had no emesis and who used no rescue drugs.
Time Frame: 24-72 hours
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Group | SyB D-0701: Low Dose Group | SyB D-0701: High Dose Group
Number analyzed (Participants) | 56 | 59 | 60
Percentage of participants
  First irraditation | 91.1 | 91.5 | 98.3
  Second irradiation | 94.5 | 96.5 | 98.3
  Third irradiation | 92.7 | 98.2 | 100.0
Statistical Analysis 1: Comparison: Placebo Group vs SyB D-0701: Low Dose Group; Statistical analysis for complete response rate after the first irradiation; Test type: Superiority or Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Placebo Group vs SyB D-0701: High Dose Group; Statistical analysis for complete response rate after the first irradiation; Test type: Superiority or Other; p = 0.1051, Fisher Exact
Statistical Analysis 3: Comparison: Placebo Group vs SyB D-0701: Low Dose Group; Statistical analysis for complete response rate after the second irradiation; Test type: Superiority or Other; p = 0.6761, Fisher Exact
Statistical Analysis 4: Comparison: Placebo Group vs SyB D-0701: High Dose Group; Statistical analysis for complete response rate after the second irradiation; Test type: Superiority or Other; p = 0.3513, Fisher Exact
Statistical Analysis 5: Comparison: Placebo Group vs SyB D-0701: Low Dose Group; Statistical analysis for complete response rate after the third irradiation; Test type: Superiority or Other; p = 0.2060, Fisher Exact
Statistical Analysis 6: Comparison: Placebo Group vs SyB D-0701: High Dose Group; Statistical analysis for complete response rate after the third irradiation; Test type: Superiority or Other; p = 0.0511, Fisher Exact

7. Secondary Outcome: Adverse Events
Description: Adverse event is any untoward medical occurrence experienced by a subject irrespective of causal relationship with the study drug, and includes the unexpected signs, clinically significant fluctuations of laboratory data, and aggravation of disease, symptoms or complications. Adverse events are coded using the preferred terms (PT) of Medical Dictionary for Regulatory Activities (MedDRA) version 15.0.
Time Frame: Up to 192 hours
Population: Safety population:
  The safety population consisted of all subjects enrolled, except for subjects with Good Clinical Practice (GCP) non-compliance and those who failed to receive the study treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo Group | SyB D-0701: Low Dose Group | SyB D-0701: High Dose Group
Number analyzed (Participants) | 60 | 63 | 62
Participants
  Number of subjects with any adverse event | 51 | 55 | 45
  Number of subjects with adverse drug reaction | 14 | 17 | 16
  Number of subjects with SAE | 1 | 0 | 0
  Number of death | 0 | 0 | 0

8. Secondary Outcome: Severe (Grade 3 or More) Adverse Events
Description: The severity of AEs were graded on a 5-point scale (Grade 1 to 5) according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
  Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe or medically significant but not immediately life-threatening, Grade 4: Life-threatening consequences, Grade 5: Death related to AE
Time Frame: Up to 192 hours
Population: Safety population:
  The safety population consisted of all subjects enrolled, except for subjects with GCP non-compliance and those who failed to receive the study treatment.
Measure: Number; unit: Number of events
Arm/Group | Placebo Group | SyB D-0701: Low Dose Group | SyB D-0701: High Dose Group
Number analyzed (Participants) | 60 | 63 | 62
Number of events
  Grade 3 : lymphopenia | 0 | 1 | 0
  Grade 3 : nausea | 2 | 0 | 0
  Grade 3 : urethritis | 0 | 1 | 0
  Grade 3 : lymph node abscess | 1 | 0 | 0
  Grade 3 : blood pressure increased | 0 | 1 | 0
  Grade 3 : C-reactive protein increased | 1 | 0 | 0
  Grade 3 : lymphocyte count decreased | 3 | 7 | 3
  Grade 3 : neutrophil count increased | 1 | 0 | 0
  Grade 3 : white blood cell count decreased | 3 | 0 | 0
  Grade 3 : blood alkaline phosphatase increased | 0 | 0 | 1
  Grade 3 : hyponatraemia | 0 | 1 | 0
  Grade 3 : decreased appetite | 1 | 0 | 0
  Grade 3 : rash maculo-papular | 0 | 1 | 0
  Grade 4 : lymphocyte count decreased | 1 | 0 | 0

9. Secondary Outcome: Skin Manifestations at Study Drug Application Site
Description: The investigator or sub-investigator recorded skin manifestations observed after removal of the study drug.
  Skin manifestations were counted for each type of patches (placebo patch, SyB D-0701 15 cm2 patch, SyB D-0701 25 cm2 patch).
Time Frame: Up to 192 hours
Population: Skin manifestations were counted for each type of patch applied to the subjects in the safety population.
  * Placebo patch : 60-1+63+60=182 (One subject in placebo group did not applied 15 cm2 patch.)
  * SyB D-0701 15 cm2 patch : 62
  * SyB D-0701 25 cm2 patch : 62+63=125
Measure: Number; unit: Number of events
Groups:
- Placebo Patch: Placebo 15 cm2 patch was applied to subjects in placebo group and low dose group.
  Placebo 25 cm2 patch was applied to subjects in placebo group.
- SyB D-0701 15 cm2 Patch: SyB D-0701 15 cm2 patch (11.25 mg) was applied to subjects in high dose group.
- SyB D-0701 25 cm2 Patch: SyB D-0701 25 cm2 patch (18.75 mg) was applied to subjects in low dose group and high dose group.
Arm/Group | Placebo Patch | SyB D-0701 15 cm2 Patch | SyB D-0701 25 cm2 Patch
Number analyzed (Participants) | 182 | 62 | 125
Number of events
  Skin manifestations: reacted | 15 | 7 | 14
  Clearly identifiable erythema | 12 | 5 | 12
  Erythema + papules | 3 | 2 | 2
  Erythema + papules + small blisters | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 192 hours
Description: The safety population was used in the analysis of adverse events. The safety population consisted of all subjects enrolled, except for subjects with GCP non-compliance and those who failed to receive the study treatment.
Groups:
- SyB D-0701: Low Dose Group: Study drug patches [Low dose group (18.75 mg): SyB D-0701 15 cm2 placebo patch + SyB D-0701 25 cm2 patch (18.75mg)] assigned at the Case Registration Center are applied to either the right or left upper arm at 12 to 24 hours prior to the start of radiotherapy and left as is until 24 hours after completion of the third irradiation.
Arm/Group | Placebo Group | SyB D-0701: Low Dose Group | SyB D-0701: High Dose Group
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/63 | 0/62
Other Adverse Events (participants affected / at risk) | 51/60 | 55/63 | 45/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Group (N=60) | SyB D-0701: Low Dose Group (N=63) | SyB D-0701: High Dose Group (N=62)
Lymph node abscess (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Group (N=60) | SyB D-0701: Low Dose Group (N=63) | SyB D-0701: High Dose Group (N=62)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 4 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 3 | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 14 | 7
Diarrhoea (Gastrointestinal disorders) | 9 | 6 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 10 | 8 | 9
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0
Application site dermatitis (General disorders) | 1 | 0 | 0
Application site erythema (General disorders) | 6 | 9 | 9
Application site pruritus (General disorders) | 9 | 5 | 10
Application site rash (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 2 | 2 | 2
Oedema peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Application site vesicles (General disorders) | 0 | 1 | 0
Application site papules (General disorders) | 1 | 1 | 2
Application site swelling (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Urethritis (Infections and infestations) | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radiation associated pain (Injury, poisoning and procedural complications) | 3 | 1 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Glucose urine present (Investigations) | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 30 | 33 | 29
Neutrophil count decreased (Investigations) | 3 | 2 | 3
Neutrophil count increased (Investigations) | 2 | 1 | 0
Platelet count decreased (Investigations) | 2 | 0 | 0
Protein total decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 16 | 13 | 14
White blood cell count increased (Investigations) | 2 | 1 | 0
Platelet count increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 2
Blood pressure increased (Investigations) | 1 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results without prior approval from the sponsor.